CLINICAL TRIAL: NCT00354692
Title: A Randomized Cross-over Pilot Study of the Effect of Sodium Ferric Gluconate Complex vs. Iron Sucrose on Proteinuria in Non-dialysis Chronic Kidney Disease Patients
Brief Title: Effect of Two Iron Preparations on Protein in the Urine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FER0601
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Kidney Failure, Chronic; Anemia, Iron-Deficiency
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia, Iron-Deficiency | interventions — ferric gluconate; Ferric Oxide, Saccharated

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Sodium Ferric Gluconate and Iron sucrose

INTERVENTIONS:
Drug: Sodium Ferric Gluconate and Iron sucrose

SUMMARY:
This pilot study will compare the effects of sodium ferric gluconate complex and iron sucrose on urine concentrations of various chemicals including protein

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe anemia
* Iron deficiency
* Moderate to severe chronic kidney disease
* Age ≥ 18 or greater and able to give informed consent

Exclusion Criteria:

* Receiving dialysis
* Known sensitivity to Sodium Ferric Gluconate Complex in Sucrose Injection, Iron sucrose USP, or any of their components
* Clinically unstable
* Indication of iron sufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in urine protein | 180 minutes

SECONDARY OUTCOMES:
Change in various urine chemicals | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adel R. Rizkala, Pharm.D., MS, Study Director — Watson Laboratories, Inc.
Locations (2):
- United States (2):
  - Glendale, California
  - Shreveport, Louisiana

REFERENCES:
- [Result] Agarwal R, Rizkala AR, Kaskas MO, Minasian R, Trout JR. Iron sucrose causes greater proteinuria than ferric gluconate in non-dialysis chronic kidney disease. Kidney Int. 2007 Sep;72(5):638-42. doi: 10.1038/sj.ki.5002422. Epub 2007 Jul 11. PMID 17622274